CLINICAL TRIAL: NCT01023425
Title: Comparative Assessment of Clinical Efficacy of Donepezil Between the Naive Group and the Switching Group
Brief Title: Clinical Trial of Donepezil Between the Naive Group and the Switching Group
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: Eisai Korea Inc. (Industry)
Responsible Party: Principal Investigator, Doh Kwan Kim, Professor, Samsung Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008-02-072
Record Dates: First submitted 2009-11-30; First posted 2009-12-02 (Estimated); Last update posted 2016-01-06 (Estimated); Status verified 2016-01

CONDITIONS: Alzheimer's Disease; Dementia
Keywords: naive group; switching group; treatment response; Efficacy; Adverse event
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — Donepezil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- switching group (Experimental): switching patients with Alzheimer's disease(AD) from galantamine or rivastigmine to donepezil because they were not responding adequately
  Interventions: Drug: donepezil
- naive group (Experimental): naive patients with AD who initiated therapy with donepezil
  Interventions: Drug: donepezil

INTERVENTIONS:
Drug: donepezil — from 5mg to 10mg, once a day, 12 months
  Other Names: donepezil-aricept

SUMMARY:
To compare the clinical efficacy of donepezil between the naive group and the switching group.

DETAILED DESCRIPTION:
The purposes of this study are:

1. to compare the efficacy between switching patients with Alzheimer's disease (AD) from galantamine or rivastigmine to donepezil because they were not responding adequately, and naive patients with AD who initiated therapy with donepezil
2. to help to clinicians in choosing the best treatment

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of probable AD according to the criteria of the NINCDS-ADRDA
2. Korean version Mini-Mental State Examination scores between 10 and 26
3. History of cognitive decline that had been gradual in onset and progressive over at least 6 months
4. A caregiver who could assist the patient with medication, attend the assessment and provide information about the patient.

Exclusion Criteria:

1. they had evidence of any neurodegenerative diseases other than AD (i.e. Parkinson's disease, Huntington's disease)
2. Psychiatric disorder or severe behavioral disturbances that required psychotropic medications
3. Cerebral injuries induced by trauma, hypoxia, and/or ischemia
4. Clinically active cerebrovascular disease; History of seizure disorder
5. Other physical conditions that required acute treatment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2008-02; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Alzheimer's Disease Assessment Scale-Cognitive, Korean version (ADAS-Cog-K) | 13 weeks, 26 weeks, 39 weeks, 52 weeks

SECONDARY OUTCOMES:
Seoul Activities of Daily Living (S-ADL) | 13 weeks, 26 weeks, 39 weeks, 52 weeks
Seoul-Instrumental Activities of Daily Living (S-IADL) | 13 weeks, 26 weeks, 39 weeks, 52 weeks
Korean Neuropsychiatric Inventory (K-NPI) | 13 weeks, 26 weeks, 39 weeks, 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Doh Kwan Kim, PhD, M.D., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea